CLINICAL TRIAL: NCT01352858
Title: Phase 1 Study of Autologous Tolerogenic Dendritic Cells for Rheumatoid Arthritis
Brief Title: Autologous Tolerogenic Dendritic Cells for Rheumatoid Arthritis (AutoDECRA)
Acronym: AutoDECRA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Arthritis Research UK (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AutoDECRA 1.0
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis; RA; Auto-immune disorders
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Arthroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TolDC (Experimental): Experimental arm - TolDC administered arthroscopically
  Interventions: Drug: TolDC
- Control (Placebo Comparator): Arthroscopy & saline irrigation alone
  Interventions: Drug: Arthroscopy & saline irrigation alone

INTERVENTIONS:
Drug: TolDC — Tolerogenic dendritic cells (TolDC), derived ex vivo from autologous monocytes, administered arthroscopically into an inflamed knee following saline irrigation.
  Arms: TolDC
Drug: Arthroscopy & saline irrigation alone
  Arms: Control

SUMMARY:
This is a study which will look at safety, feasibility and acceptability of a new therapy called tolerogenic dendritic cells (TolDC), derived from the patient's own white blood cells, which will be injected into the knee joints of rheumatoid arthritis patients, using a procedure called arthroscopy (a camera examination of a joint). The investigators are also looking to see if the drug has any effect on the disease activity (if it can help in RA) and whether the drug can affect the immune system. The investigators aim to treat 12 patients in total, 9 with TolDC and 3 with a control treatment. Three doses of TolDC will be tested, 3 patients per dose. Subjects will have RA and at least one swollen knee joint. They will undergo a knee ultrasound scan, fill in a series of questionnaires, have their knee aspirated (fluid taken out) and finally undergo a procedure called leukapheresis (removal of white blood cells) from which the treatment will be manufactured. Subsequently they will undergo 3 arthroscopies (camera examination of the knee joint) over a period of about 12 weeks. On the first arthroscopy they will have the TolDC injected into their knee joint. They will then spend the night at the Clinical Research facility for observation. Over the next 5 days they will be telephoned daily by the study doctor to check how they are, and will be reassessed if needed. About 2 weeks later they will have their second arthroscopy to look for effects of treatment, and the third will take place at 13 weeks (end of study) or sooner if the knee appears to get worse.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent and to comply with the study protocol
* At least 6 month's disease duration
* ACR Functional Class I-III
* Age 18 years or over
* Active disease, including an inflamed (native) knee joint
* Failure (or intolerance of) at least one disease modifying anti-rheumatic drug (DMARD), including current therapy
* Morning stiffness in the target joint ≥ 30 minutes
* Willing and able to undergo arthroscopic procedures under local anaesthetic
* Stable dose of non-steroidal anti-inflammatory drug (NSAID) or corticosteroid (prednisolone≤10mg) for ≥4 weeks
* No intramuscular glucocorticoid administration for ≥ 6 weeks
* Stable dose of disease-modifying anti-rheumatic drug (DMARD) for ≥8 weeks

Exclusion Criteria:

* Use of other investigational medicinal products within 30 days prior to study entry (defined as date of recruitment into study)
* Patients who have received rituximab therapy and whose B-cell count remains below the normal range. Patients who have received any other cell depleting therapies and whose cell counts have not returned to the normal range, at the discretion of the principal investigator.
* Serious or unstable co-morbidity deemed unsuitable by PI, eg. COPD, cardiac failure
* History of malignancy (except treated basal cell carcinoma of skin)
* Known active infection at screening visit or at baseline (except fungal nail infection)
* Infection requiring hospitalization or IV antibiotics within 6 weeks of baseline
* Immunization with live vaccine within 6 weeks of baseline
* History of recurrent or chronic infection
* History of hepatitis B or C, syphilis, HIV or HTLV-1/2 infections
* Injection of target joint with glucocorticoids within 6 weeks of baseline
* Hb<10g/dL; neutrophils< 2.00 x109/L; platelets <150x109/L; ALT/ALP>2x upper limit of normal; elevated serum creatinine at screening visit.
* Major surgery within 8 weeks of baseline or planned within 3 months from baseline
* Pregnancy, or women planning to become pregnant within the study period, or women who are breast feeding
* Females or males of child bearing potential unwilling to use adequate contraception for duration of study
* Patients taking anticoagulants
* Known hypersensitivity to local or systemic corticosteroid therapy or local anaesthetic.
* Poor venous access or medical condition precluding leukapheresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-02; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
The proportion of patients experiencing AEs and SAEs following the intra-articular administration of TolDC. | within 3 months of injection

SECONDARY OUTCOMES:
• The proportion of RA patients who enter the study, from whom GMP-grade TolDC of sufficient quality can be prepared (the success rate of the TolDC preparation procedure). | Within one week of donation of blood for extraction of TolDC
• The proportion of patients who grade the trial and its related procedures as acceptable. | At final study visit, 3 months after study intervention.
  Trial participants will assess acceptability of study specific procedures via an 'acceptability questionnaire' administered at the last study visit
Systemic RA disease activity | At baseline and at 7, 14 and 91 days post intervention
  Disease Activity Score using 28 joints (DAS28)
Knee function | At baseline and at 7, 14 and 91 days post-intervention
  Function will be assessed using the Health Assessment Questionnaire (HAQ), a standard instrument used in RA

CONTACTS AND LOCATIONS:
Locations (1):
- Newcastle University, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Bell GM, Anderson AE, Diboll J, Reece R, Eltherington O, Harry RA, Fouweather T, MacDonald C, Chadwick T, McColl E, Dunn J, Dickinson AM, Hilkens CM, Isaacs JD. Autologous tolerogenic dendritic cells for rheumatoid and inflammatory arthritis. Ann Rheum Dis. 2017 Jan;76(1):227-234. doi: 10.1136/annrheumdis-2015-208456. Epub 2016 Apr 26. PMID 27117700